CLINICAL TRIAL: NCT01949623
Title: Biomarkers In Retinitis Pigmentosa (BIRP)
Acronym: BIRP
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: BIRP
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Retinitis Pigmentosa
Keywords: RP
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Paracentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anterior Chamber fluid from the eye
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RP patients: Retinitis Pigmentosa patients
  Interventions: Other: Anterior Chamber (AC) tap
- Controls: Patients who will be undergoing surgery for macular hole, epiretinal membrane, or vitreomacular traction, patients who have a retinal detachment , patients with neovascular age related macular degeneration and patients with diabetic retinopathy.
  Interventions: Other: Anterior Chamber (AC) tap

INTERVENTIONS:
Other: Anterior Chamber (AC) tap — Aqueous Samples will be collected for measurement of biomarkers

SUMMARY:
In this study, markers of oxidative stress will be measured in the aqueous humour and plasma of RP patients compared to controls.

DETAILED DESCRIPTION:
People with Retinitis Pigmentosa have loss of night vision followed by loss of central vision due to damage and death of photoreceptors. One of the mechanisms causing damage is high levels of oxygen in the eye. This damage produces specific biomarkers which can be measured. In this study, these biomarkers will be assessed in people with Retinitis Pigmentosa and compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age more than or equal to 18 years
* For the study group, patients diagnosed with Retinitis Pigmentosa by the investigators
* For the control group, patients undergoing vitreoretinal surgery for macular hole, epiretinal membrane, vitreomacular traction, retinal detachment, neovascular Age-related Macular Degeneration (AMD) and Diabetic Retinopathy will be eligible

Exclusion Criteria:

* Patients with active or suspected ocular or periocular infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinitis Pigmentosa patients and Controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Aqueous levels of markers of oxidative stress in patients with RP and controls. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No